CLINICAL TRIAL: NCT01394523
Title: A Prospective, Double-blinded, Randomized Comparison of Caudal Analgesia Versus Ultrasound Guided Rectus Sheath Blocks for Umbilical Herniorrhaphy in the Pediatric Population
Brief Title: Caudal Versus Rectus Sheath Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interim power analysis was prohibitive to continuing the study
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tarun Bhalla, MD, Attending Anesthesiologist, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB11-00363
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Umbilical Hernia
MeSH Terms: conditions — Hernia, Umbilical | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Caudal epidural (Active Comparator): The caudal epidural block will be delivered with 1.5ml/kg of 0.25% Bupivacaine up to a maximum of 30 mL.
  Interventions: Drug: Bupivacaine
- Rectus sheath (Active Comparator): The rectus sheath block will be performed with 0.1ml/kg of 0.25% Bupivacaine on each side at the T9-T10 distribution under ultrasound guidance.
  Interventions: Drug: Bupivacaine
- Local (Active Comparator): The surgeon will inject either 0.5% Bupivicaine 0.5ml/kg or 0.25% Bupivicaine 1ml/kg at the surgeon's discretion.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 0.25% or 0.5%

SUMMARY:
The literature has clearly demonstrated that the effective treatment of postoperative pain in infants and children is challenging. In an effort to improve postoperative analgesia while limiting opioid-related adverse effects, there continues to be an increased use of regional anesthetic techniques in infants and children. Although the pediatric caudal remains the most commonly used pediatric regional anesthetic technique, it has been demonstrated that effective analgesia can be provided with the use of peripheral nerve blockade even in the pediatric-aged patient. The purpose of this study is to prospectively compare post-operative pain relief in pediatric patients undergoing umbilical hernia repair who have received either a caudal block or bilateral rectus sheath blocks for analgesia

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Weight less than or equal to 20 kg
* Presenting for repair of umbilical hernia

Exclusion Criteria:

* ASA physical status > II
* Weight greater than 20 kg
* Co-morbid diseases (cardiac, pulmonary, neurological disease)
* Patients having concomitant procedures (circumcision, orchiopexy, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caudal Epidural: The caudal epidural block was delivered with 1.5ml/kg of 0.25% Bupivacaine up to a maximum of 30 mL.
  Bupivacaine: 0.25% or 0.5%
- Rectus Sheath: The rectus sheath block was performed with 0.1ml/kg of 0.25% Bupivacaine on each side at the T9-T10 distribution under ultrasound guidance.
  Bupivacaine: 0.25% or 0.5%
- Local: The surgeon injected either 0.5% Bupivicaine 0.5ml/kg or 0.25% Bupivicaine 1ml/kg at the surgeon's discretion.
  Bupivacaine: 0.25% or 0.5%
Period: Overall Study
Arm/Group | Caudal Epidural | Rectus Sheath | Local
Started | 13 | 13 | 13
Completed | 12 | 13 | 13
Not Completed | 1 | 0 | 0
Not completed — Unable to place block | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caudal Epidural | Rectus Sheath | Local | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.2 (1.5) | 4.3 (1.6) | 4.6 (1.2) | 4.4 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 6 | 22
  Male | 7 | 3 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Score
Description: Hannallah et al developed the Objective Pain Scale (OPS) to monitor pain in children after surgery. Parameters: (1) systolic blood pressure, (2) crying, (3) movement, (4) agitation (confused, excited), (5) complains of pain (may not be possible in younger children). Interpretation: minimum score: 0; maximum score: 10; maximum score if too young to complain of pain: 8; the higher the score, the greater the degree of pain.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: pain score
Arm/Group | Caudal Epidural | Rectus Sheath | Local
Number analyzed (Participants) | 12 | 13 | 13
pain score | 2.9 (3.3) | 3.1 (3.1) | 2.1 (2.7)

ADVERSE EVENTS:
Arm/Group | Caudal Epidural | Rectus Sheath | Local
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes